CLINICAL TRIAL: NCT04177576
Title: Evaluation of New Biomarkers of Thrombosis in Myeloproliferative Neoplasms
Acronym: MPN-BIOCLOT
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2018/50
Record Dates: First submitted 2019-10-30; First posted 2019-11-26 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-10

CONDITIONS: Myeloproliferative Neoplasm
Keywords: Polycythemia Vera (PV); Essential Thrombocythemia (ET); Neutrophil Extracellular Trap (NET); Thrombosis
MeSH Terms: conditions — Myeloproliferative Disorders; Polycythemia Vera; Thrombocythemia, Essential; Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma aliquots
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with myeloproliferative neoplasms (MPN): Patients diagnosed with Polycythemia Vera (PV) or Essential Thrombocythemia (ET)
  Interventions: Biological: 2 additional tubes of blood

INTERVENTIONS:
Biological: 2 additional tubes of blood — 2 additional tubes of blood will be collected to prepare plasma aliquots used tomeasure markers of neutrophil activation

SUMMARY:
Thrombosis is the main cause of morbidity and mortality in patients with myeloproliferative neoplasms (MPN). However, the pathogenesis of thrombosis in MPN is still largely elusive. Neutrophils can release their decondensed chromatin as a network of extracellular fibers named NET for "neutrophils extracellular trap". NETs are known to be procoagulant. Our main objective is to quantify NETs biomarkers expression in MPN patients and define if they could be used as prognostic factors in the outcome of thrombosis in these patients.

DETAILED DESCRIPTION:
Myeloproliferative neoplasms (MPN) are acquired clonal hematopoietic stem cell disorders, characterized by an increase in one or more myeloid lineages. The Philadelphia chromosome negative (Ph-) MPN include polycythemia vera (PV) with an excess of red blood cells, essential thrombocythemia (ET) with an increase in platelets and primary myelofibrosis (PMF). Arterial and venous thromboses are the main causes of morbidity and mortality in MPN with reported incidences ranging from 12-39% in PV and 11-25% in ET. The pathogenesis of thrombosis in MPN patients is complex and still largely elusive. The overproduction of neutrophils could be an important risk factor in the thrombus formation. Indeed neutrophils are known to promote thrombosis when they release their decondensed chromatin as a network of extracellular fibers named NET for "neutrophils extracellular trap". Increased NETosis has been reported in a mouse model of MPN. The main objective of this study is to investigate whether NET biomarkers are associated with increased thrombotic risk in patients with ET. Indeed, an international thrombotic prognostic score has been published in ET, ie the IPSET Thrombosis score (history of thrombosis, age, presence of JAK2V617F, cardiovascular risk factors).

Plasma from MPN patients will be collected, at the time of diagnosis, and measure markers of neutrophil activation, including NET biomarkers. The IPSET Thrombosis score will be evaluated in patients with ET and the correlation between the IPSET Thrombosis score and these biomarkers will be measured.

No follow-up is required for this study.

ELIGIBILITY:
Inclusion Criteria:

* Adults (age ≥18 years),
* Patients diagnosed with Polycythemia vera (PV) or essential thrombocythemia (ET) according to WHO 2008 criteria,
* Affiliated to the national social security system,
* Signed informed consent form will be required for each included subject after having read the information note,
* Patient agreeing to be included in the FIMBANK register and having signed the corresponding consent

Exclusion Criteria:

* Adults (age >18 years), male or female,
* Patients treated with heparin or undergoing cytoreductive treatment,
* Pregnant or lactating woman,
* Person under guardianship, tutorship or other legal protection scheme or incapable of giving consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with myeloproliferative neoplasms (MPN), diagnosed with Polycythemia vera (PV) or essential thrombocythemia (ET)
Sampling Method: Non-Probability Sample
Enrollment: 397 (Actual)
Dates: Start 2020-02-24 (Actual); Primary Completion 2022-01-26 (Actual); Study Completion 2022-01-26 (Actual)

PRIMARY OUTCOMES:
Correlation between NET biomarkers and the risk of thrombosis | 1 day
  Correlation between NET biomarkers measurated in plasma samples and the risk of thrombosis evaluated by the prognostic score IPSET thrombosis

SECONDARY OUTCOMES:
Correlation between MPO-DNA levels (measured by absorbance at 405 nm) and a history of thrombosis | 1 day
Correlation between MPO-DNA levels (measured by absorbance at 405 nm) and the subtype of MPN disease (ET or PV) | 1 day
Correlation between MPO-DNA levels (measured by absorbance at 405 nm) and the presence of JAK2V617F mutation | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Chloé JAMES, Principal Investigator — University Hospital, Bordeaux
Locations (24):
- France (24):
  - CHU Angers, Angers
  - CH Annecy Genevois, Annecy
  - CH Avignon, Avignon
  - CHU Bordeaux, Hématologie Biologique, Bordeaux
  - CHU Bordeaux, Hématologie Clinique et Thérapie Cellulaire, Bordeaux
  - CHU Bordeaux, Médecine Interne, Bordeaux
  - Institut Bergonié, Bordeaux
  - CHRU Brest, Brest
  - CHU Henri Mondor - APHP, Créteil
  - CH Dax, Dax
  - CHU Dijon, Dijon
  - CHU Limoges, Limoges
  - Centre Léon Bérard, Lyon
  - CH Mont de Marsan, Mont-de-Marsan
  - CHU Nancy, Nancy
  - Hôpital Européen Georges Pompidou - APHP, Paris
  - Hôpital Saint-Louis - APHP, Paris
  - CH Perpignan, Perpignan
  - CHU Poitiers, Poitiers
  - CH Rochefort, Rochefort
  - CH Roubaix, Roubaix
  - IUCT-Oncopôle, Toulouse
  - CH Valenciennes, Valenciennes
  - Hôpital Paul Brousse, Villejuif

IPD SHARING:
Plan to Share IPD: No